CLINICAL TRIAL: NCT01659502
Title: Investigator's Initiated Phase II Study for Pancreatic Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tiltan Pharma Ltd. (Industry)
Responsible Party: Principal Investigator, Tzivia Berkman, Dr Ayala Hubert, Tiltan Pharma Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLH-207
Record Dates: First submitted 2012-07-23; First posted 2012-08-07 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Pancreatic Cancer
Keywords: Patients
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — TL-118

ARMS (1):
- TL-118 alone or with pancreas cancer chemotherapy (Experimental)
  Interventions: Drug: TL-118

INTERVENTIONS:
Drug: TL-118 — TL-118 investigational product is supplied as an oral liquid for daily administration at a specific dosing regimen. Treatment protocol includes weekly therapy cycles

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of TL-118 alone or in combination with pancreatic cancer chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years at enrollment.
2. Locally Advanced Pancreatic Cancer and/or Metastatic Pancreatic Cancer which failed to respond to one or two lines of chemotherapy
3. The patient has histologically or cytologically confirmed pancreatic cancer.
4. Patient has measurable disease by radiological imaging techniques as defined according to Response Evaluation Criteria in Solid Tumors (RECIST).
5. ECOG performance status ≤ 2
6. Adequate renal function.
7. Adequate hepatic function
8. Adequate bone marrow reserve -
9. Resolution of prior therapy acute adverse events.
10. Patient is capable of swallowing.
11. Patient's Informed Consent.

Exclusion Criteria:

1. Hypersensitivity to one or more of the TL-118 active components
2. Known Glucose-6-phosphate-dehydrogenase deficiency (G6PD).
3. Known CNS or Brain metastases
4. Patient has received 3 or more different prior chemotherapies for the treatment of pancreatic cancer
5. Any significant change in treatment within the 14 days before screening or an un-stable medical condition that may affect patient participation or evaluation in the study.
6. Concurrent use of any other investigational product or within 28 days before study entry.
7. Chronic treatment with: (a) immunosuppressive agent other than systemic corticosteroid, (b) patients who are under chronic treatment with NSAIDs with the exception of Aspirin at a daily dose ≤ 100mg.
8. Use of supplements or complementary medicines/botanicals, except for conventional multivitamin supplements, calcium, selenium and soy supplements.
9. Patients at increased risk of gastro intestinal bleeding such as patients with known active gastro intestinal ulcer, erosive gastritis or varices, as confirmed by gastroscopy performed within one year before screening.
10. Serious or uncontrolled co-existent diseases that are likely to significantly increase the risks associated with TL-118 therapy (e.g. severe cardiovascular disease, congestive heart failure, recent myocardial infarction, significant vascular disease, active or uncontrolled autoimmune disease, active or uncontrolled infection).
11. Patient has known historical or active infection with HIV, hepatitis B, or hepatitis C
12. Serious or non-healing wound, ulcer or bone fracture.
13. Circumstances likely to interfere with absorption of orally administrated drugs.
14. History of noncompliance to medical regimens or coexisting conditions precluding full compliance with study protocol, or any other condition that in the discretion of the Investigator may preclude safe and complete study participation.
15. Subjects unwilling or unable to comply with study protocol.
16. Know pregnancy or breast-feeding women.
17. Women of child bearing potential not exercising two methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Measurement | Baseline up to 2 years
  Clinical Benefit Measurement is a composite of measurements of pain (analgesic consumption and pain intensity), performance status and weight. Clinical benefit requires an improvement in at least one parameter, without worsening in any others, sustained for at least 4 weeks

SECONDARY OUTCOMES:
Safety and tolerability | Baseline up to 2 years
  Safety and tolerability profiles will be judged by:
  * Local and systemic toxicities.
  * Number, type and degree of toxicities as measured by the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) v4.0
Response Rate (RR) | RR measured every 8 weeks after enrollment up to 2 years
Overall Survival | OS measured at 16 and 52 weeks after treatment initiation or at death, whichever comes first up to 2 years
Progression Free Survival (PFS) | PFS measured at 8 weeks after enrollment until the date of first documented progression or date of death, whichever comes first, up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel